CLINICAL TRIAL: NCT05645003
Title: Effect of Repetative Transcranial Magnetic Stimulation Therapy on Neuropathic Pain in Patients With Spinal Cord Injury
Brief Title: Transcranial Magnetic Stimulation Therapy in Neuropathic Painful Spinal Cord Injury Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Nuran Eyvaz, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMSSKY2022
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain; Neurological Diseases or Conditions
Keywords: Repetitive Transcranial Magnetic Stimulation; Neurological Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-frequency real-time rTMS protocol (Experimental): It was planned to apply a total of 1200 beats to the dorsolateral prefrontal cortex daily at a frequency of 10 HZ at 110% intensity of the motor threshold for 15 sessions.
  Interventions: Device: High-frequency real-time rTMS protocol
- Sham rTMS Protocol (Sham Comparator): It was planned to apply daily sham rTMS to the dorsolateral prefrontal cortex for 15 sessions.
  Interventions: Device: Sham rTMS Protocol

INTERVENTIONS:
Device: High-frequency real-time rTMS protocol — It was planned to apply a total of 1200 beats to the dorsolateral prefrontal cortex daily for 15 sessions. Along with the daily rTMS session, patients will continue to use the drugs in the medical treatment (pregabalin, gabapentin, carbamazepine) at the same effective dose. No dose changes will be made during rTMS sessions.
  Arms: High-frequency real-time rTMS protocol
Device: Sham rTMS Protocol — It was planned to apply a to the dorsolateral prefrontal cortex daily for 15 sessions. Along with the daily rTMS session, patients will continue to use the drugs in the medical treatment (pregabalin, gabapentin, carbamazepine) at the same effective dose. No dose changes will be made during rTMS sessions.
  Arms: Sham rTMS Protocol

SUMMARY:
The aim of our study is to investigate the effect of high-frequency Repetitive Transcranial Magnetic Stimulation(rTMS) therapy applied to the dorsolateral PFC (DLPFC) area on neuropathic pain in patients with spinal cord injury. In this area, there are very few studies on the effectiveness of rTMS treatment added to medical treatment in neuropathic pain. In addition, the number of studies comparing the effect of rTMS therapy applied to the DLFPC area is very few.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is associated with widespread disability due to its detrimental effects on various bodily functions. Neuropathic pain is one of the most challenging complications after SCI and can have a significant impact on daily life.

There are supportive criteria for the diagnosis of neuropathic pain associated with SCI: onset of pain within one year after SCI, absence of primary association between pain with movement, inflammation or other local tissue damage, burning, tingling, pins and needles, throbbing pain, squeezing pain, Detection of 1 or more of the pain descriptors such as freezing pain, allodynia or hyperalgesia within the pain distribution support neuropathic pain due to spinal cord injury.

Pharmacological and interventional treatments are often tried in the treatment of neuropathic pain, but their success is often limited. Another option that has been used as an innovative approach in the treatment of neuropathic pain in recent years is pain regulation with rTMS. As one of the non-invasive brain stimulation techniques, rTMS is suggested to be useful in the treatment of central neuropathic pain. While most studies to date have mainly targeted the primary motor cortex (M1), which is contralateral to the pain side, fewer studies have reported analgesic effects after stimulation of other cortical areas such as the dorsolateral PFC (DLPFC). The analgesic mechanisms of rTMS to the DLPFC are thought to be through the same mechanism as stimulation of the M1 motor cortex.

The aim of our study; To investigate the effect of high frequency rTMS applications on patients with SCI on their neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 20-70, who applied to the AFSU Physical Medicine and Rehabilitation inpatient service with the diagnosis of spinal cord injury and

* Having spinal cord injury with neurophatic pain at least six months ago,
* Able to follow two-stage verbal commands,
* Agreeing to participate in the study voluntarily and regularly,
* Patients who are medically stable (no previous myocardial infarction, no musculoskeletal problems) will be included in our study.

Exclusion Criteria:

Having an important comorbid disease such as severe heart disease (aortic stenosis, angina, hypertrophic cardiomyopathy, arrhythmia, pacemaker) and uncontrolled hypertension,

* Epilepsy,
* History of antiepileptic drug use,
* Intracranial metal object,
* Presence of in-ear implant,
* Cognitive dysfunction,
* Lower extremity peripheral nerve injury,
* With malignancy and active infection,
* Infection on the skin in the application area,
* Having an open wound,
* Having inflammatory disease,
* Orthopedic injuries that can limit maximum effort contractions,
* Having a brain lesion or a history of drug use that will affect the seizure threshold,
* Patients with increased intracranial pressure or uncontrolled migraine will not be included.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Visual Analog Scale (VAS) at 15 day and 6 week. | up to 6 week
  It is evaluated between 0-10. 10 means severe pain, 0 means no pain. Night and day VAS assessment will be questioned.

SECONDARY OUTCOMES:
Change from baseline The Leeds Assessment of Neuropathic Symptoms & Signs Pain Scale(LANSS) at 15 day and 6 week. | up to 6 week
  LANSS consists of two parts; The first part, filled out by the patient himself, and the second part, which includes the doctor's brief physical examination.If score < 12, neuropathic mechanisms are unlikely to be contributing to the patient's pain.If score≥ 12, neuropathic mechanisms are likely to be contributing to the patient's pain.
Change from baseline Short form McGill Pain questionnaire(SF-MPQ) at 15 day and 6 week. | up to 6 week
  It is evaluated between 0-45. It is an expanded version of the abbreviated McGill Questionnaire by adding 7 new items specific to neuropathic pain.The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Change from baseline Short form 36 (SF-36) at 15 day and 6 week. | up to 6 week
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score was between 0 ( disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.
Change from baseline Beck Depression Scale at 15 day and 6 week. | up to 6 week
  It is a self-assessment scale that can be used in healthy patient groups to determine the risk of depression in the individual and to measure the level and severity of depressive symptoms. It includes a total of 21 self-assessment questions. It provides a four-point Likert-type measurement. Each item gets progressively increasing points between 0 and 3, and the total score is obtained by summing them up. The total score ranges from 0 to 63. 0-9: indicates minimal depression, 10-18: indicates mild depression, 19-29: indicates moderate depression, 30-63: indicates severe depression. Higher total scores indicate more severe depressive symptoms.
Beck Anxiety Scale at 15 day and 6 week. | up to 6 week
  It is a self-assessment scale that can be used in healthy patient groups to measure the frequency of anxiety experienced by the individual. It includes a total of 21 self-assessment questions. It provides a four-point Likert-type measurement. Each item gets progressively increasing points between 0 and 3, and the total score is obtained by summing them up. The total score ranges from 0 to 63. 8-15 is considered mild anxiety, 16-25 moderate anxiety, 26-63 severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Background] Nardone R, Holler Y, Langthaler PB, Lochner P, Golaszewski S, Schwenker K, Brigo F, Trinka E. rTMS of the prefrontal cortex has analgesic effects on neuropathic pain in subjects with spinal cord injury. Spinal Cord. 2017 Jan;55(1):20-25. doi: 10.1038/sc.2016.87. Epub 2016 May 31. PMID 27241450
- [Background] Yang QH, Zhang YH, Du SH, Wang YC, Fang Y, Wang XQ. Non-invasive Brain Stimulation for Central Neuropathic Pain. Front Mol Neurosci. 2022 May 19;15:879909. doi: 10.3389/fnmol.2022.879909. eCollection 2022. PMID 35663263
- [Background] Li L, Huang H, Yu Y, Jia Y, Liu Z, Shi X, Wang F, Zhang T. Non-invasive Brain Stimulation for Neuropathic Pain After Spinal Cord Injury: A Systematic Review and Network Meta-Analysis. Front Neurosci. 2022 Feb 11;15:800560. doi: 10.3389/fnins.2021.800560. eCollection 2021. PMID 35221889